CLINICAL TRIAL: NCT00916682
Title: Structure and Function of Salivary Proteins
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Tufts University (Other); Boston University (Other); Boston Medical Center (Other); University of North Carolina, Chapel Hill (Other); Ahura Scientific, Inc. (Industry)
Responsible Party: Ahmet Uluer, DO, Children's Hospital, Boston
Other Study IDs: X07-03-0142
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cystic Fibrosis

SUMMARY:
This study seeks to provide point-of-care clinical diagnostic systems for the diagnosis of current disease status using saliva as a sample specimen.

DETAILED DESCRIPTION:
The overall hypothesis of this study is that whole saliva and its components, due to its direct anatomic relation to the airways, provides a window on the composition and nature of the disease-specific response in the bronchial, sinus, and nasal airways. By examining proteins created in saliva, we hope to validate that saliva is an important diagnostic tool for for rapid analysis of respiratory status. We further propose that rapid salivary diagnostics will improve patient care in prevalent respiratory diseases with frequent health care utilization and high morbidity, such as asthma, chronic obstructive pulmonary disease (COPD), and cystic fibrosis (CF).

ELIGIBILITY:
Inclusion Criteria:

* 6 or more years of age
* confirmed Cystic Fibrosis

Exclusion Criteria:

* Pregnant

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be approached during their pulmonary clinic appointment or while they are inpatient at Children's Hospital, Boston.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Uluer, DO, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hosptital, Boston, Boston, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://ase.tufts.edu/chemistry/walt/saliva/